CLINICAL TRIAL: NCT07013851
Title: Phase II Clinical Trial to Assess the Efficacy of Dostarlimab as Neoadjuvant Therapy in Patients With MMRd/MSI-H Stage II-III Endometrial Cancer
Brief Title: Clinical Trial to Assess the Efficacy of Dostarlimab as Neoadjuvant Therapy in Patients With MMRd/MSI-H Stage II-III Endometrial Cancer
Acronym: NADIA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICO 137-E; 2024-512021-81-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-28; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: MMRd/MSI-H Stage II-III Endometrial Cancer
MeSH Terms: interventions — dostarlimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Patients will be treated in the neoadjuvant setting with dostarlima 500 mg (30') every 3 weeks for 4 cycles.All participants will undergo surgery within 6 weeks following the final dose of neoadjuvant dostarlimab. After surgery, adjuvant chemotherapy, including dostarlimab, will be administered as follows:
  Stage II EC:
  VBT/EBRT (completed within >14 weeks after surgery) + Adjuvant dostarlimab 1000 mg Q6W x 9 cycles (54 weeks total).
  Stage III EC:
  1. Concurrent EBRT+cisplatin followed by carboplatin + paclitaxel OR
  2. Sequential: EBRT followed by carboplatin + paclitaxel OR
  3. Chemotherapy alone: carboplatin + paclitaxel
     * Adjuvant dostarlimab 500 mg Q3W x 4-6 cycles (in combination with chemotherapy) plus 1000 mg Q6W x 6-7 cycles (54 weeks total).
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — Patients will be treated in the neoadjuvant setting with dostarlima 500 mg (30') every 3 weeks for 4 cycles.All participants will undergo surgery within 6 weeks following the final dose of neoadjuvant dostarlimab. After surgery, adjuvant chemotherapy, including dostarlimab, will be administered as follows:
  Stage II EC:
  VBT/EBRT (completed within >14 weeks after surgery) + Adjuvant dostarlimab 1000 mg Q6W x 9 cycles (54 weeks total).
  Stage III EC:
  1. Concurrent EBRT+cisplatin followed by carboplatin + paclitaxel OR
  2. Sequential: EBRT followed by carboplatin + paclitaxel OR
  3. Chemotherapy alone: carboplatin + paclitaxel
     * Adjuvant dostarlimab 500 mg Q3W x 4-6 cycles (in combination with chemotherapy) plus 1000 mg Q6W x 6-7 cycles (54 weeks total).

SUMMARY:
The study for which participation is requested is a phase II clinical trial to assess the efficacy of dostarlimab as neoadjuvant therapy in patients with MMRd/MSI-H stage II-III endometrial cancer. The study is conducted in Spain with an estimated number of 25 patients for phase II. The main objective of this phase-II study is to evaluate the clinical complete response (cCR) after neoadjuvant therapy with dostarlimab.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects at least 18 years of age, who are able to understand the study procedures and agree to participate in the study by providing written informed consent.
2. Histologically confirmed new diagnosis of endometrial adenocarcinoma (endometrioid subtype only) by central pathology review.
3. MMRd status confirmed by IHC by central laboratory.
4. Subject must provide adequate tumor tissue sample at screening for MMR/MSI status testing. The quality of the tumor tissue sample must be confirmed by the central laboratory during screening.
5. Subjects must have primary stage II or III (FIGO 2023) disease. Pelvic involvement is included. Stage IIIB2 patients with metastasis to pelvic peritoneum are excluded.
6. ECOG performance status of 0 or 1.
7. Treatment naïve patients without previous radiation or systemic therapy, including hormonal therapy.
8. Participants should have adequate organ function defined as:

   * ANC ≥1.5×109/L
   * Hemoglobin ≥9 g/dL ≥5.6 mmol/L
   * Platelets ≥100×109/L
   * AST and ALT ≤2.5×ULN
   * Bilirubin ≤1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
   * For patients not taking anticoagulant: INR ≤ 1.5x or PT ≤1.5× ULN. Activated partial thromboplastin time (aPTT) ≤1.5× ULN. Participants receiving anticoagulants PT or PTT are within therapeutic range of intended use of anticoagulants.
   * Renal function parameters of GFR ≥30 mL/min/1.73m2 (institutional creatinine ≤1.5×ULN) Note: Blood count test should be performed without transfusion or receipt of colony stimulating factors within 4 weeks prior to obtaining the blood sample.
9. Contraceptive use by subjects should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

   * The participant is a woman of nonchildbearing potential OR
   * The participant is a woman of childbearing potential, using a contraceptive method that is highly effective (with a failure rate of <1% per year) during the study treatment period and for at least 120 days after the last dose of study treatment and agrees not to donate eggs (ova or oocytes) for the purpose of reproduction during this period.

Exclusion Criteria:

1. Diagnosis of clear cell, serous, undifferentiated or carcinosarcoma or other uterine mesenchymal tumor such as endometrial stromal sarcoma, leiomyosarcoma, or other types of sarcomas. Adenosarcomas and neuroendocrine tumors are not allowed either.
2. Any previous radiation or systemic therapy.
3. ECOG performance status ≥2.
4. Immunodeficiency or treatment with chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy.
5. Subject has a concomitant malignancy, or a prior non-endometrial invasive malignancy who has been disease-free for <3 years or who received any active treatment in the last 3 years for that malignancy. Non-melanoma skin cancer is allowed.
6. Participants have current active or history of pneumonitis or interstitial lung disease.
7. Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
8. Participant has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.
9. Immunocompromised patients are not allowed.
10. Allergy: Participant cannot have history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies or fusion proteins, sensitivity to any of the study treatments or components thereof, or a history of drug or other allergy that contraindicates their participation.
11. Participant has experienced any of the following with prior immunotherapy: any immune-related AE (irAE) of Grade 3 or higher, immune-related severe neurologic events of any grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain-Barré syndrome, or transverse myelitis), exfoliative dermatitis of any grade (SJS, TEN, or DRESS syndrome), or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary.
12. Participant has clinically significant cardiovascular disease within 6 months of enrolment.
13. Prohibited medications: Participant has received systemic steroid therapy (>10 mg daily prednisone or equivalent) within 7 days before the first dose of the study treatment or is receiving any other form of immunosuppressive medication. Replacement therapy (adrenal or pituitary insufficiency) is not considered a form of systemic therapy. Use of inhaled corticosteroids, local steroid injection, or steroid eye drops is allowed.
14. Subject has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both.
15. Subject has known active hepatitis B. Participants who are HBsAg positive are eligible if they have undetectable HBV viral load prior to enrolment.
16. Subject has a positive HCV antibody test result at Screening or within 3 months prior to first dose of study intervention. NOTE: Participants with a positive HCV antibody test result due to prior resolved disease can be enrolled, only if a confirmatory negative HCV RNA test is obtained.
17. Subject has a positive HCV RNA test result at Screening or within 3 months prior to first dose of study intervention. NOTE: The HCV RNA test is optional and participants with negative HCV antibody test are not required to undergo HCV RNA testing as well.
18. Participants with known HIV infection are allowed with the following requirements:

    * Documented evidence of plasma HIV-1 RNA persistently <50 copies/mL ≤3 months prior to AND at Screening. In the >3 to 12 months prior to Screening, plasma HIV-1 RNA consistently <50 c/mL required; if single increases ≥50 c/mL occurred, they cannot have been persistent nor associated with antiretroviral resistance per investigator assessment AND
    * CD4 cell count >350 cells/mm3 over past 12 months and at Screening (and no measurement ≤350 cells/mm3 during that time period) AND
    * Must be on an uninterrupted combination antiretroviral therapy regimen for at least 3 months prior to Screening, with combination antiretroviral therapy regimen consistent with locally recommended guidelines.
    * Participants with history of CDC Stage 3 AIDS-defining disease (CDC, 2014; also known as acquired immunodeficiency syndrome - defining disease) are allowed if AIDS-defining disease has been treated and cured or is stable for ≥3 months prior to study entry. Cutaneous Kaposi's sarcoma not requiring systemic therapy is allowed.
    * No history of HIV-associated non-Hodgkin lymphoma ≤5 years prior to study entry.
    * No treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
19. Subject has not recovered adequately (Grade ≤1) from AEs and/or complications from any major surgery prior to starting therapy.
20. Subject has a known intolerance or hypersensitivity to dostarlimab active substance, infused protein products, or any of its excipients.
21. Subject is currently participating and receiving study treatment or has participated in a study of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment.
22. Subject is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active infection requiring systemic therapy.
23. Subject has received, or is scheduled to receive, a live vaccine within 30 days before first dose of study treatment, during study treatment, and for up to 180 days after receiving the last dose of study treatment.
24. Participant is pregnant or breastfeeding.
25. Participant has received a live vaccine within 30 days of planned start of study therapy. COVID-19 vaccines that do not contain live viruses are allowed. Note: mRNA and adenoviral-based COVID-19 vaccines are considered non-live.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical complete response (cCR) after neoadjuvant dostarlimab. | 43 months
  cCR: Efficacy measured by the proportion of patients who had cCR after neoadjuvant dostarlimab. cCR is defined as the absence of tumor persistence evaluated by MRI, CT, PET scan, pelvic exam, and review of surgical specimen.

SECONDARY OUTCOMES:
To evaluate the pathologic complete response (pCR) after neoadjuvant dostarlimab. | 51 months
  pCR: Efficacy measured by the proportion of patients who had pCR having undergone surgery after neoadjuvant dostarlimab. pCR is defined as the absence of invasive tumor in the surgical specimen by local pathology review.
To evaluate the overall response rate (ORR) of neoadjuvant dostarlimab. | 51 months
  ORR: Efficacy measured by ORR, which is defined as the number of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of response evaluable patients (according to RECIST v1.1).
To evaluate disease-free survival (DFS). | 51 months
  DFS: Efficacy measured by DFS, which is defined as the time in months from date of dostarlimab's first dose to date of local or distant recurrence (assessed radiologically by the investigator or by histopathologic confirmation), or death due to any cause, whichever occurs first.
To evaluate the median of overall survival (mOS). | 51 months
  mOS: Efficacy measured by mOS, which is defined as the median of time in months from date of dostarlimab's first dose to date of death due to any cause. OS will be censored on the last date a patient was known to be alive.
To evaluate the safety and tolerability of dostarlimab in the neoadjuvant setting. | 51 months
  Toxicity will be assessed by adverse events related to study drugs, detected through physical examinations and laboratory tests, and graded according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Español de Investigación en Cáncer Ginecológico (GEICO), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No